CLINICAL TRIAL: NCT03155685
Title: Of the Use of Antipsychotics in Palliative Care : Prospective, Multicenter, Observational Study.
Brief Title: Use of Antipsychotics in Palliative Care (NEUROPAL)
Acronym: NEUROPAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 16-151
Record Dates: First submitted 2017-05-05; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Antipsychotics in Palliative Care
Keywords: antipsychotic; palliative care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are not lots of recommendations for the use of antipsychotics in palliative care. The National Agency for Accreditation and Evaluation in Health (ANAES) and the French Society for Accompaniment and Palliative Care, in 2002, make it the first-line treatment for confusion in palliative care, but there are no information on the molecules to be used, the dosage or the route of administration.

Many symptoms can motivate the prescription of an antipsychotic and many molecules exist. Their mode of action is substantially the same but their pharmacological properties sometimes give them different beneficial effects or side effects. They are studied in psychiatry but very little in palliative care.

Depending on the symptom (s) presented by the patient, either of these antipsychotics may be preferred. Use appear to differ from one center to another.

The investigator propose a multicenter, prospective, observational study describing the antipsychotics used according to the symptom.

This study should include 100 patients over the age of 18 years in palliative care (regardless of pathology) who are not taking antipsychotics and for whom the decision to introduce an antipsychotic is made regardless of the symptom.

The purpose of this work is to describe the most commonly used antipsychotic according to a particular symptom, as well as the dosage and route of administration.

The investigator will also evaluate the 7-day efficacy of the chosen antipsychotic on the symptom that motivated the prescription, and we will compare the dosages of the associated treatments before and after the introduction of this new treatment.

DETAILED DESCRIPTION:
The investigator will question the practice of palliative care physicians in several centers regarding the use of antipsychotics.

When a patient meeting the inclusion criteria has been identified by an investigating physician. The participant fills out a questionnaire containing some general information about the investigating physician and the patient, followed by a first questionnaire, called A Form (to be completed on D0, when the antipsychotic is introduced) with 8 questions on the prescribing symptom, antipsychotic used and associated therapies.

Seven days later, the same physician will fill out a second form, called B Form (to be completed on D7), with 9 questions on treatment efficacy, possible modifications and associated treatments.

Each investigating physician includes a maximum of 4 patients over the 6-month inclusion period.

Once the 4 questionnaires have been completed (Form A and Form B), he / she returns it to the principal investigator of the study, by e-mail to etudeneuropal@gmail.com, or by mail: Dr Marie LEPOUPET, Mobile Pain-Palliative Care Unit CHU, Côte de Nacre Avenue, 14,000 CAEN.

ELIGIBILITY:
Inclusion Criteria:

* all patients over the age of 18 years in palliative care, regardless of the stage of their illness, and according to the definition used by ANAES and SFAP (all patients suffering from a serious, progressive disease involving life-threatening, advanced or terminal).
* having a social security cover
* not taking antipsychotics at the time of inclusion, nor within 3 days before inclusion.
* for whom the doctor, investigator, decides to prescribe an antipsychotic, whatever it is, whatever the symptom motivating this prescription, whatever the dosage and the route of administration used.

Drugs related to antipsychotics, such as metoclopramide, metopimazine, alizapride or domperidone, are not included in this study.

Exclusion Criteria:

* patients with contraindications to antipsychotics
* patients already taking an antipsychotic, or for whom an antipsychotic was stopped less than 3 days ago.
* patients under 18 years of age.
* pregnant women
* patients protected by the law
* patients who are unable to refrain from participating in a study, and for whom the entourage (a trusted person, relatives, etc.) is also unable to refrain from such participation.

The study can be released at any time at the request of the patient and / or his entourage.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in palliative care, regardless of the stage of their progressive, life-threatening disease (as defined by ANAES and SFAP)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
antipsychotic name (ICD) | when the antipsychotic is first prescribed by the investigator and so the patient included in the study, up to 6 months between the beginning of the study and the patient inclusion
  name (ICD) of the antipsychotic used according to the symptom presented by the patient
administration route | when the antipsychotic is first prescribed by the investigator and so the patient included in the study, up to 6 months between the beginning of the study and the patient inclusion
  Per os, Subcutaneous, Intravenous, Sublingual, Intramuscular
daily dosage | when the antipsychotic is first prescribed by the investigator and so the patient included in the study, up to 6 months between the beginning of the study and the patient inclusion
  milligrams per day

SECONDARY OUTCOMES:
simple verbal scale of efficiency of the antipsychotic on the symptom | evaluation by the patient or the investigator if patient impossible, 7 days after the introduction of the antipsychotic.
  simple verbal scale : weak, medium, strong, very strong
change of dosage of the associated treatments | comparison between the dosage of each associated treatment at Day 0 and Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Christophe KASSEL, Study Director — University Hospital, Caen

IPD SHARING:
Plan to Share IPD: No